CLINICAL TRIAL: NCT00116103
Title: A Phase II, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of Tacrolimus Inhalation Aerosol in Subjects With Persistent Asthma
Brief Title: A Study of the Safety and Efficacy of Tacrolimus Inhalation Aerosol in Subjects With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-0-213
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Asthma
Keywords: Treatment Effectiveness; Treatment Efficacy; Investigational, Therapies; Asthma; Antiasthmatics; Antiasthmatic agents
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: Tacrolimus Inhalation Aerosol

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of tacrolimus inhalation aerosol in subjects with persistent asthma.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind, placebo-controlled, parallel-group, multi-center designed trial is to determine the safety and efficacy of tacrolimus inhalation aerosol in subjects with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of persistent asthma for at least 6 months
* Require use of beta-agonists at least four times per week

Exclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease (COPD)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-06; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in FEV1 from baseline to end-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Medical Monitor, MD, Study Director — Astellas Pharma US, Inc.
Locations (21):
- United States (21):
  - Scottsdale, Arizona
  - Encinitas, California
  - Los Angeles, California
  - San Diego, California
  - San Jose, California
  - Denver, Colorado
  - Daytona Beach, Florida
  - Miami, Florida
  - Boise, Idaho
  - River Forest, Illinois
  - South Bend, Indiana
  - St Louis, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Providence, Rhode Island
  - Spartanburg, South Carolina
  - San Antonio, Texas
  - Madison, Wisconsin
  - Milwaukee, Wisconsin